CLINICAL TRIAL: NCT00002184
Title: A Phase II, Stratified, Randomized, Double-Blind, Multi-Center Study of the Safety and Efficacy of Adefovir Dipivoxil (ADF) at Two Dose Levels in Triple Combination Therapies With Protease Inhibitors (PI) and Nucleoside Reverse Transcriptase Inhibitors (RTI) for the Treatment of HIV-Infected Patients With CD4 Cell Counts >= 100/mm3 and HIV-1 RNA Copy Numbers >= 5,000 Copies/Ml and Prior RTI Therapy But No Prior PI Therapy
Brief Title: A Phase II, Stratified, Randomized, Double-Blind, Multi-Center Study of the Safety and Efficacy of Adefovir Dipivoxil (ADF) at Two Dose Levels in Triple Combination Therapies With Protease Inhibitors (PI) and Nucleoside Reverse Transcriptase Inhibitors (RTI) for the Treatment of HIV-Infected Patient
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 232E
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-10

CONDITIONS: HIV Infections
Keywords: HIV-1; Dose-Response Relationship, Drug; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Zidovudine; Stavudine; HIV Protease Inhibitors; CD4 Lymphocyte Count; Lamivudine; RNA, Viral; Saquinavir; Nelfinavir; Reverse Transcriptase Inhibitors; Adenine; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Nelfinavir; Carnitine; adefovir dipivoxil; Saquinavir; Lamivudine; Stavudine; Zidovudine

INTERVENTIONS:
Drug: Nelfinavir mesylate
Drug: Levocarnitine
Drug: Adefovir dipivoxil
Drug: Saquinavir
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine

SUMMARY:
To evaluate the safety and tolerance of the combination of adefovir dipivoxil at two comparative doses and nelfinavir plus saquinavir SGC administered orally (Group 1) vs. the combination of adefovir dipivoxil and nelfinavir plus either zidovudine, lamivudine, or stavudine (Group 2) vs. the combination of adefovir dipivoxil and saquinavir SGC plus either zidovudine, lamivudine, or stavudine (Group 3) in HIV-infected patients with prior nucleoside reverse transcriptase inhibitor therapy but no prior exposure to protease inhibitors who have CD4 cell counts >= 100 cells/mm3 and an HIV-1 RNA baseline copy number >= 5000 copies/ml. To determine the proportion of patients whose plasma HIV-1 RNA level falls below the level of detection (<500 copies/ml) at 20 weeks of study therapy and the average reduction in HIV-1 RNA from baseline through study week 20. To evaluate the durability of the antiviral response through 48 weeks of study in patients who continue on study therapy after week 24.

DETAILED DESCRIPTION:
This protocol is a stratified, randomized, double-blind, dose-comparative study of the safety and efficacy of adefovir dipivoxil in combination with nelfinavir and saquinavir soft gel capsules (SGC) or adefovir dipivoxil in combination with nelfinavir or saquinavir SGC plus a nucleoside analog (zidovudine, lamivudine, or stavudine).

Patients will be randomized to adefovir dipivoxil with nelfinavir and saquinavir or adefovir dipivoxil with nelfinavir or saquinavir plus a nucleoside analog (zidovudine, lamivudine, or stavudine). Within each treatment arm, patients will be randomized to 1 of 2 doses of adefovir dipivoxil in a blinded manner. Patients randomized to receive a nucleoside analog will then be assigned to receive either zidovudine, lamivudine, or stavudine based upon their previous RTI therapy. A daily dose of L-carnitine will be administered to all patients.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Laboratory diagnosis of HIV infection (positive HIV antibody test confirmed by Western blot, p24 antigen assay, HIV-1 RNA, or HIV-1 culture).
* An HIV-1 RNA plasma titer >= 5000 copies/ml within 14-21 days prior to the baseline visit.
* CD4 cell count >= 100 cells/mm3 within 14-21 days prior to the baseline visit.
* A minimum life expectancy of at least 1 year.
* Signed, informed consent from parent or legal guardian for those patients < 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms and conditions are excluded:

* Active, serious infections (other than HIV infection) requiring parenteral antibiotic or antiviral therapy. Patients will be considered recovered from such infectious episodes if at least 2 weeks elapsed following the cessation of parenteral therapy before the baseline visit.
* Exhibiting evidence of a gastrointestinal malabsorption syndrome or chronic nausea or vomiting that may confer an inability to receive an orally administered medication.
* Malignancy other than cutaneous Kaposi's sarcoma (KS) or basal cell carcinoma. Patients with biopsy-confirmed cutaneous KS are eligible, but must not have received any systemic therapy for KS within 4 weeks prior to baseline and are not anticipated to require systemic therapy during the study.
* Any other clinical condition that in the opinion of the investigator would make the patient unsuitable for study or unable to comply with the dosing requirements.

Patients with any of the following prior conditions are excluded:

* A new AIDS-defining event diagnosed within 1 month prior to baseline.
* Significant history of peripheral neuropathy.

  1. Treatment with immunomodulating agents such as systemic corticosteroids, IL-2, or interferons.
* Ritonavir, indinavir, nevirapine, delavirdine, didanosine, dideoxycytidine, interferon alpha, interferon beta, isoniazid, rifampin, investigational agents (except upon Sponsor approval), chemotherapeutic agents (systemic), terfenadine, astemizole, cisapride, triazolam, and midazolam.

  1. Prior use of adefovir dipivoxil.
* Prior use of any antiretroviral protease inhibitor.
* Immunizations within 30 days of baseline.
* Antiretroviral vaccine therapy within 60 days of baseline.
* Treatment in the 4 weeks prior to baseline with immunomodulating agents such as systemic corticosteroids, IL-2, or interferons.
* Any other investigational drug within 30 days prior to baseline.
* Any prior therapy that, in the opinion of the investigator, would make the patient unsuitable for study or unable to comply with the dosing requirements.

Required:

Prior therapy for > 4 weeks with any licensed nucleoside analog inhibitor of HIV reverse transcriptase.

Patients with current alcohol or substance abuse judged by the investigator to potentially interfere with patient compliance.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120

CONTACTS AND LOCATIONS:
Locations (15):
- United States (13):
  - Phoenix Body Positive, Phoenix, Arizona
  - Krauss Med Partners / Dept of Research and Development, Los Angeles, California
  - UCLA Care Ctr, Los Angeles, California
  - Davies Med Ctr, San Francisco, California
  - Blick Med Associates, Greenwich, Connecticut
  - George Washington Med Ctr, Washington D.C., District of Columbia
  - Johns Hopkins Univ School of Medicine, Baltimore, Maryland
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - North Shore Community Hosp, Manhassett, New York
  - Associates of Med and Mental Health, Tulsa, Oklahoma
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Mem Hosp of Rhode Island, Pawtucket, Rhode Island
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
- Puerto Rico (2):
  - Hosp Regional de Ponce - Area Vieja, Ponce
  - San Juan AIDS Program, Santruce